CLINICAL TRIAL: NCT06908759
Title: Risk of Falling Assessment in a Population of Patients With Cardiovascular Diseases Undergoing Cardiac Rehabilitation
Brief Title: Risk of Falling and Cardiac Rehabilitation
Acronym: CARDIO-BALANCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 119/SR/24
Record Dates: First submitted 2025-03-26; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Risk of Falling; Elderly (People Aged 65 or More); Cardiovascular Diseases
Keywords: risk of fall; cardiac rehabilitation
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Exercise; Dosage Forms

STUDY DESIGN:
Intervention Model Description: The study will enroll 150 patients of both sexes with known cardiac disease, referred to the cardiac rehabilitation unit of IRCCS San Raffaele of Rome following an acute cardiac event requiring hospitalization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- supervised exercise in cardiac rehabilitation (Experimental): group 1: patients will perform supervised exercise training in the gym of San Raffaele IRCCS of Rome
  Interventions: Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION
- home-based exercise (Active Comparator): group 1: patients will be asked to perform not supervised exercise training at home according to european guidelines for people with cardiovascular diseases
  Interventions: Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION

INTERVENTIONS:
Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION — In the first phase of the study all enrolled patients will perform exercise in the context of an in-hospital intesive rehabilitation after the acute event. At discharge they will be randomized in two groups: supervised exercise in the context of a cardiac rehabilitation facility or home-based exercise

SUMMARY:
Background and Rationale Cardiac rehabilitation (CR) is a key intervention for patients with chronic heart disease or recent acute cardiovascular events. In elderly and frail patients, CR aims not only to improve functional capacity but also to maintain or recover independence in daily activities. Hospitalization following an acute event often leads to bed rest, which-even after just 2-3 days-can cause hypokinetic syndrome, characterized by loss of muscle tone, orthostatic hypotension, decreased mobility, and psychological decline, including depression. Moreover, immobility increases thrombotic risk and vascular complications.

To mitigate these effects, CR is initiated promptly after clinical stabilization and includes three phases:

1. Phase I - In-hospital rehabilitation
2. Phase II - Early outpatient rehabilitation
3. Phase III - Long-term maintenance Elderly patients are particularly vulnerable to falls due to the combined effects of reduced muscle strength, orthostatic hypotension, cognitive decline, and pre-existing sarcopenia-often exacerbated by acute events and immobility. Approximately 60% of cardiac patients hospitalized for acute events present with moderate-to-high fall risk. Fall risk in this population is multifactorial, involving cardiovascular issues (e.g., arrhythmias, orthostatic hypotension), medication effects, and non-cardiac factors such as vision loss, balance impairment, neuromuscular conditions, and cognitive deficits.

DETAILED DESCRIPTION:
Cardiac rehabilitation is recommended for patients with chronic heart diseases and those who have experienced a recent acute cardiovascular event. Among the main goals of cardiac rehabilitation following an acute event is the recovery of functional capacity or, alternatively-especially in elderly and frail individuals-the maintenance or recovery of autonomy, at least in activities of daily living, within the limits imposed by the cardiac impairment.

An acute cardiovascular event requiring hospitalization is often accompanied by a period of varying duration of immobility and bed rest. Bed rest lasting more than 2-3 days may lead to a hypokinetic syndrome characterized by reduced or absent movement autonomy, loss of muscle tone, orthostatic hypotension (deconditioning), and often a decline in mood that may progress to depression. Furthermore, immobility is associated with increased thrombotic risk and consequently a greater chance of vascular complications.

To counteract bed rest and its complications, cardiac rehabilitation is initiated as soon as the patient's condition stabilizes and includes three phases:

* Phase I rehabilitation (in-hospital)
* Phase II rehabilitation (early outpatient)
* Phase III rehabilitation (maintenance phase) [1]. Loss of muscle mass and tone, orthostatic hypotension, and cognitive impairments all contribute to an increased fall risk in the elderly. It is estimated that approximately 60% of heart disease patients hospitalized for an acute event have a medium-to-high fall risk [2,3].

Specifically in cardiac patients, multiple additional factors may contribute to fall risk in this population, including:

1. Cardiovascular conditions:

   * These may cause sudden reductions in cardiac output and/or inadequate increases in peripheral resistance, resulting in pre-syncope or syncope.
   * These include:

     1. Tachyarrhythmias or bradyarrhythmias (sustained ventricular tachycardia; severe bradycardia; advanced sinoatrial or atrioventricular block).
     2. Orthostatic hypotension: Often caused by autonomic dysfunction related to prolonged bed rest and/or use of blood pressure-lowering medications such as vasodilators. Excessive reduction in blood volume from diuretics can also contribute.
2. Non-cardiac conditions:

   * Cardiac patients, especially older ones, may have reduced vision, balance disorders, cognitive impairments, or neuromuscular disorders that make walking unstable.
   * Additionally, elderly cardiac patients-particularly those with heart failure-have a high prevalence of sarcopenia. This condition, often present at baseline, may be significantly worsened by the acute clinical event and resulting hypo-/immobility.

Study Objectives

* Primary objective: To evaluate the effect of cardiac rehabilitation on fall risk in elderly cardiac patients following a recent acute event requiring hospitalization.

  o We hypothesize that patients completing a supervised rehabilitation cycle will score better on the Conley Scale than those discharged directly home.
* Secondary endpoints include:

  * Effects of rehabilitation on balance in elderly cardiac patients
  * Effects of rehabilitation on sleep quality, anxiety, and stress levels
  * The impact of rehabilitation will also be evaluated based on hospital stay duration and total volume of physical training performed

ELIGIBILITY:
Inclusion Criteria:

- Age > 65 years

Recent acute cardiac event, including:

1. Cardiac surgery (CABG, aortic and/or mitral valve replacement, mitral valvuloplasty, or combined CABG + valve surgery)
2. Recent myocardial infarction treated with percutaneous revascularization
3. Episode of acute heart failure

Exclusion Criteria:

Persistent clinical instability, defined as:

* Marked hypotension (BP ≤ 95/60 mmHg) or hypertension (BP ≥ 160/100 mmHg)
* Bradycardia (HR < 50 bpm) or tachycardia (HR > 115 bpm)
* Resting dyspnea
* Signs and symptoms of infection

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of cardiac rehabilitation on the risk of falling in elderly cardiac patients following a recent acute event requiring hospitalization. | Fron enrollment to the end of the in-hospital phase and after 12 weeks from discharge
  The risk of falling will be assessed through the Conley scale. We will consider the percentage changes in the score obtained in the Conley scale at different evaluation times in relation to the study design

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCs San Raffaele, Rome, RM, Italy